CLINICAL TRIAL: NCT03477591
Title: McMaster Choices Study: Evaluating the Impact of Evidence-based Information About PSA Testing on Prostate Cancer Screening Decisions
Brief Title: Evaluating the Impact of Evidence-based Information About PSA Testing on Prostate Cancer Screening Decisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 4351
Record Dates: First submitted 2018-03-12; First posted 2018-03-26 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
Keywords: Screening; PSA testing; Patient Decision Aid
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Evidence + PDA (Experimental): Evidence-based information on PSA testing such as blog posts, plain language evidence summaries and web resource ratings (quality-appraised online resources), plus a blog post on PDAs and the relevant decision aid from the Portal database
  Interventions: Other: Evidence-based information; Other: Patient Decision Aid
- Evidence only (Experimental): The same evidence-based information as group 1 (Evidence + PDA), but without the PDA to quantify the effect of accessing evidence through the Portal alone
  Interventions: Other: Evidence-based information
- Attention control (Sham Comparator): Information on how to distinguish high from low-quality health information, not specific to cancer screening or PDAs
  Interventions: Other: Sham information

INTERVENTIONS:
Other: Evidence-based information — Evidence-based information on PSA testing such as blog posts, plain language evidence summaries and web resource ratings (quality-appraised online resources).
  Arms: Evidence + PDA; Evidence only
Other: Patient Decision Aid — Patient Decision Aid for prostate cancer screening decision
  Arms: Evidence + PDA
Other: Sham information — Educational information not specific to PSA testing or cancer screening
  Arms: Attention control

SUMMARY:
Patient decision aids are tools that help guide individuals through a healthcare-related decision making process. They help users combine evidence-based information and recommendations by a health care provider with their personal needs, values and preferences. Through this project, Dr. Dobbins and her research team will explore whether the use of patient decision aids with high-quality and user-friendly summaries of research evidence, or summaries of research evidence alone, help to improve the quality of decision making by men facing prostate cancer screening decisions.

DETAILED DESCRIPTION:
Guidelines for prostate screening in Canada are based on low-moderate quality evidence of effectiveness and screening is associated with potential harms. Patient Decision Aids (PDAs) are tools that assist users to understand treatment options, risks and benefits to align decisions with values and preferences. The investigators would now like to know whether use of a PDA alongside evidence-based information provided through the McMaster Optimal Aging Portal, or simply access to evidence-based information alone, can help users to make informed decisions about prostate cancer screening in men.

ELIGIBILITY:
Inclusion Criteria:

* English speaking men, > 50 years old

Exclusion Criteria:

* History of prostate cancer or PSA test in the last 12 months

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | Change from baseline to 6-mo
  Decisional Conflict Scale

SECONDARY OUTCOMES:
Decision quality | Change from baseline to 6-mo
  Decision Quality Worksheet for PSA testing
Preparation for decision making | Change from baseline to 6-mo
  Preparation for decision making scale
Screening behaviour | Change from baseline to 6-mo
  Congruency between self-reported screening status and stated decision

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Dobbins, RN, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No